CLINICAL TRIAL: NCT04185623
Title: Time Lag for Oocyte Denudation:Is it a Better Choice for ICSI Outcome?!
Brief Title: Time Lag for Oocyte Denudation: A Better Choice for ICSI Outcome?!
Status: Completed | Type: Observational
Sponsor: Ahmed Saad (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Sponsor-Investigator, Ahmed Saad, Assistant professor of Obstetrics & Gynecology, Benha University
Organization: Benha University (Other)
Other Study IDs: Hawaa-8
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female
Keywords: denudation timing ICSI timing oocyte aging
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (immediate denudation): Oocytes were denudated immediately after oocyte retrieval and were microinjected at 4 hours from ovum pickup. Microinjection was performed on all matured oocytes only and they were cultured to blastocyst stage.The rates of maturation, fertilization, good quality blastulation, chemical pregnancy and clinical pregnancy were analysed and compared between the two groups.
  Interventions: Procedure: denudation time lag
- Group B ( 2hs denudation after ovum pickup): Oocytes were denudated 2 hours after retrieval and were microinjected at 4 hours from ovum pickup. Microinjection was performed on all matured oocytes only and they were cultured to blastocyst stage.The rates of maturation, fertilization, good quality blastulation, chemical pregnancy and clinical pregnancy were analysed and compared between the two groups.
  Interventions: Procedure: denudation time lag

INTERVENTIONS:
Procedure: denudation time lag — The time between ovum pickup and denudation of oocyte

SUMMARY:
This study aiming to investigate if difference in the timing of cumulus removal post retrieval would have any critical impact on fertilization and embryonic development.

DETAILED DESCRIPTION:
Patients under 37 year old who were treated with controlled ovarian stimulation for ICSI were randomly divided into 2 groups; Group A: Oocytes were denudated immediately after oocyte retrieval , Group B: Oocytes were denudated 2 hours after retrieval and both groups were microinjected at 4 hours from ovum pickup. Microinjection was performed on all matured oocytes only and they were cultured to blastocyst stage.The rates of maturation, fertilization, good quality blastulation, chemical pregnancy and clinical pregnancy were analysed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women 24-37 years old
* With good ovarian reserve
* Induction using Long agonist protocol
* unexplained infertility

Exclusion Criteria:

* severe male factor
* Testicular samples for ICSI
* poor ovarian reserve
* no of oocytes collected less than 4

Ages: 24 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: couples who came seeking fertility through our IVF center
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Day 5, good quality blastocyst | 120 hour post ovum pickup
  Assessment were done according to gardener classification

SECONDARY OUTCOMES:
clinical pregnancy | 6 weeks from the last normal menstrual period
  Assessment was done by observation of a gestational sac at 6 wks

CONTACTS AND LOCATIONS:
Locations (1):
- Hawaa Fertility Center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after completion of the study
Supporting Information: Study Protocol, SAP
Time Frame: after 1 year for 2 months